CLINICAL TRIAL: NCT00392990
Title: A Multicenter Phase II Study Incorporating DOXIL® and Rituximab Into the Magrath Regimen for HIV-Negative and HIV-Positive Patients With Newly Diagnosed Burkitt's and Burkitt-like Lymphoma
Brief Title: Doxorubicin Hydrochloride Liposome and Rituximab With Combination Chemotherapy in Treating Patients With Newly Diagnosed Burkitt's Lymphoma or Burkitt-Like Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 06H2; P30CA060553 (NIH); NU 06H2 (Other: Northwestern University); NU-1346-018; ORTHO-NU-06H2; CDR0000509706 (Registry Identifier: PDQ); STU00004480 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma
Keywords: stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; AIDS-related peripheral/systemic lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma | interventions — OOS-A regimen; Rituximab; liposomal doxorubicin; Cyclophosphamide; Vincristine; Methotrexate; merphos; Regimen B; Ifosfamide; Etoposide; Podophyllotoxin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alternating doxil/Magrath regimen & rituximab/Magrath regimen (Experimental): Patients are stratified between high risk and low risk disease status. Low risk patients receive 3 cycles of rituximab (500 mg/m2) R-CODOX-M chemotherapy IV over 2-4 hours with intrathecal chemotherapy (Regimen A). High risk patients receive 1 cycle of R-CODOX-M chemotherapy IV followed by R-IVAC chemotherapy over 30 minutes(Regimen B); regimens A and B are then repeated.
  Interventions: Drug: Regimen A; Drug: Regimen B

INTERVENTIONS:
Drug: Regimen A — Cyclophosphamide (800 mg/m2 IV over 1 hour)+ vincristine (1.5 mg/m2 IV PUSH)+ doxorubicin (40 mg/m2 IV)+ high-dose methotrexate (2,700 mg/m2 IV over 23 hours)+ rituximab (500 mg/m2 IV)(R-CODOX-M) regimen
  Other Names: Rituximab; Doxil; pegylated liposomal doxorubicin; cyclophosphamide; Cytoxan®; CTX; CPM; Neosar®; Vincristine; Oncovin®; Vincasar PFS®; vincristine sulphate; VCR; leucocristine; LCR; Methotrexate; Methotrexate sodium; MTX; Mexate; Mexate-AQ; Folex; Folex PFS; Abitrexate; Rheumatrex; Amethopterin
Drug: Regimen B — Rituximab (500 mg/m2 IV once)+ Ifosfamide (1500 mg/m2 IV daily over 3 hours)+ Etoposide (60 mg/m2 IV daily over 1 hour), and Cytarabine (2 grams/m2 IV over 3 hours for 4 doses)
  Other Names: Rituximab; Ifosfamide; Ifex®; Etoposide; VP-16; VePesid®; VP-16-213; EPEG; epipodophyllotoxin; NSC # 141540; Cytarabine; Cytosar-U; Ara-C; Arabinosyl; cytosine arabinoside

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving rituximab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving doxorubicin hydrochloride liposome and rituximab together with combination chemotherapy works in treating patients with newly diagnosed Burkitt's lymphoma or Burkitt-like lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate (complete remission, complete remission undetermined, and partial remission) in HIV-negative or HIV-positive patients with newly diagnosed Burkitt's or Burkitt-like lymphoma treated with doxorubicin hydrochloride liposome and rituximab as part of the Magrath regimen.

Secondary

* Determine the complete remission rate in patients treated with this regimen.
* Determine progression-free and overall survival at 2 years in patients treated with this regimen.
* Determine the safety of adding rituximab to the standard Magrath regimen in these patients.
* Determine the safety of using doxorubicin hydrochloride liposome in place of doxorubicin hydrochloride in these patients.
* Determine correlative levels of rituximab and doxorubicin hydrochloride liposome in cerebrospinal fluid and peripheral blood.

OUTLINE: This is a multicenter study. Patients are stratified according to risk category (low risk vs high risk). Patients are assigned to 1 of 2 treatment regimens according to stratum.

* Regimen A (low-risk disease with no CNS involvement): Patients receive R-CODOX-M chemotherapy comprising rituximab IV over 2-4 hours on days 0 and 8; doxorubicin hydrochloride liposome IV over 30 minutes on day 1; vincristine IV on days 1 and 8; cyclophosphamide IV over 1 hour on days 1-5; and high-dose methotrexate (MTX) IV over 24 hours on day 10. Patients also receive leucovorin calcium IV beginning 36 hours after the start of MTX infusion and continuing every 6 hours until blood levels of MTX are safe. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily on days 4-8 in courses 1 and 3 and on days 6 and 7 in course 2. Beginning on day 12, daily G-CSF dosing resumes until blood counts recover. Patients receive CNS prophylaxis comprising cytarabine intrathecally (IT) on day 1 and MTX IT on day 3. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Regimen B (high-risk disease with or without CNS involvement): Patients receive R-CODOX-M chemotherapy with leucovorin calcium and G-CSF support as in regimen A for courses 1 and 3 and R-IVAC chemotherapy with leucovorin calcium and G-CSF support (as below) for courses 2 and 4. R-IVAC chemotherapy comprises high-dose ifosfamide IV over 3 hours and etoposide IV over 1 hour on days 1-5; cytarabine IV over 3 hours twice daily on days 2 and 3; and rituximab IV over 2-4 hours on day 0 and on day 6 or 7. Patients also receive leucovorin calcium orally every 6 hours on day 6 and G-CSF SC once daily beginning on day 6 or 7 and continuing until blood counts recover. Patients without CNS involvement receive CNS prophylaxis comprising cytarabine IT on days 1 and 3 and MTX IT on day 15 in courses 1 and 3 and MTX IT alone on day 5 in courses 2 and 4. Patients with proven CNS involvement at diagnosis receive cytarabine IT on days 1, 3, and 5 in course 1, on days 7 and 9 in course 2, and on days 1 and 3 in course 3. These patients also receive MTX IT on days 15 and 17 in course 1, on day 5 in courses 2 and 4, and on day 15 in course 3. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

The first 10 patients enrolled on the study undergo cerebrospinal fluid and blood collection during courses 1 and 3 for correlative biological marker and pharmacological studies.

After completion of study treatment, patients are followed at 30 days and then periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Burkitt's or Burkitt-like non-Hodgkin's lymphoma meeting 1 of the following risk criteria:

  * Low-risk disease meeting all of the following criteria:

    * Normal lactate dehydrogenase level
    * ECOG performance status 0-1
    * Ann Arbor stage I or II
    * No tumor mass over 10 cm in greatest diameter
  * High-risk disease, defined as disease not meeting low-risk criteria
* Newly diagnosed disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count ≥ 500/mm³
* Platelet count ≥ 100,000/mm³ (50,000/mm³ if bone marrow involvement is documented)
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* Bilirubin ≤ 1.5 times ULN (3 times ULN if liver metastases are present)
* Creatinine clearance > 50 mL/min
* Creatinine ≤ 2.0 mg/dL
* LVEF ≥ 45% by MUGA scan or echocardiogram
* No New York Heart Association class II-IV heart failure
* No clinically significant pericardial disease
* No myocardial infarction within the past 6 months
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No ECG evidence of acute ischemia or active conduction system abnormalities

  * Investigator must document any baseline ECG abnormality as not medically relevant
* No other malignancy within the past year except for basal cell carcinoma of the skin or in situ carcinoma of the cervix
* No other serious medical or psychiatric illness that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* Prior treatment with 1 course of any combination of rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, and/or prednisone* (CHOP)-like therapy allowed, provided the following doses are not exceeded:

  * Rituximab 750 mg/m²
  * Cyclophosphamide 1,000 mg/m²
  * Doxorubicin hydrochloride 50 mg/m²
  * Vincristine 2 mg/m²
* No other investigational drugs within the past 14 days
* No other concurrent systemic, cytotoxic, investigational, or chemotherapy agents NOTE: *No maximum dose restriction on steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02-06; Primary Completion 2011-12-03 (Actual); Study Completion 2013-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Gordon, MD, Principal Investigator — Northwestern University
Locations (8):
- United States (8):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger Cook County Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Washington University, St Louis, Missouri
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University Hospitals Case Medical Center, Cleveland, Ohio

REFERENCES:
- [Derived] Evens AM, Carson KR, Kolesar J, Nabhan C, Helenowski I, Islam N, Jovanovic B, Barr PM, Caimi PF, Gregory SA, Gordon LI. A multicenter phase II study incorporating high-dose rituximab and liposomal doxorubicin into the CODOX-M/IVAC regimen for untreated Burkitt's lymphoma. Ann Oncol. 2013 Dec;24(12):3076-81. doi: 10.1093/annonc/mdt414. Epub 2013 Oct 20. PMID 24146219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on October 4, 2006 with the first patient enrolling and starting treatment on February 6, 2007 and an accrual goal of up to 25 patients. The study was closed permanently on April 26, 2011 to further accrual with 25 patients enrolled on the study.
Pre-assignment Details: Patients were stratified as either high-risk or low-risk.
  Low Risk= patients with normal Lactic acid dehydrogenase (LDH) level, Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1, Ann Arbor stage as I or II and no tumor mass over 10 cm in greatest diameter.
  High Risk = All other patients
Groups:
- Low Risk - Treatment With 3 Cycles of R-CODOX-M: Patients are stratified between high risk and low risk disease status. Low risk patients receive 3 cycles of rituximab (500 mg/m2) R-CODOX-M chemotherapy IV over 2-4 hours with intrathecal chemotherapy (Regimen A).
  Regimen A: Cyclophosphamide (800 mg/m2 IV over 1 hour)+ vincristine (1.5 mg/m2 IV PUSH)+ doxorubicin (40 mg/m2 IV)+ high-dose methotrexate (2,700 mg/m2 IV over 23 hours)+ rituximab (500 mg/m2 IV)(R-CODOX-M) regimen
  Regimen B: Rituximab (500 mg/m2 IV once)+ Ifosfamide (1500 mg/m2 IV daily over 3 hours)+ Etoposide (60 mg/m2 IV daily over 1 hour), and Cytarabine (2 grams/m2 IV over 3 hours for 4 doses)
- High Risk - Treatment With Alternating R-CODOX-M/R-IVAC Cycles: Patients are stratified between high risk and low risk disease status.
  High risk patients receive 1 cycle of R-CODOX-M chemotherapy IV followed by R-IVAC chemotherapy over 30 minutes(Regimen B); regimens A and B are then repeated.
  Regimen A: Cyclophosphamide (800 mg/m2 IV over 1 hour)+ vincristine (1.5 mg/m2 IV PUSH)+ doxorubicin (40 mg/m2 IV)+ high-dose methotrexate (2,700 mg/m2 IV over 23 hours)+ rituximab (500 mg/m2 IV)(R-CODOX-M) regimen
  Regimen B: Rituximab (500 mg/m2 IV once)+ Ifosfamide (1500 mg/m2 IV daily over 3 hours)+ Etoposide (60 mg/m2 IV daily over 1 hour), and Cytarabine (2 grams/m2 IV over 3 hours for 4 doses)
Period: Treatment on Study
Arm/Group | Low Risk - Treatment With 3 Cycles of R-CODOX-M | High Risk - Treatment With Alternating R-CODOX-M/R-IVAC Cycles
Started | 20 | 5
Completed | 17 | 4
Not Completed | 3 | 1
Not completed — Adverse Event | 3 | 1
Period: Follow up for 2 Years
Arm/Group | Low Risk - Treatment With 3 Cycles of R-CODOX-M | High Risk - Treatment With Alternating R-CODOX-M/R-IVAC Cycles
Started (All patients that receive one dose of study drug go into the follow-up phase.) | 20 | 5
Completed | 16 | 5
Not Completed | 4 | 0
Not completed — Death | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Risk - Treated With Alternating R-CODOX-M/R-IVAC Cycles: Patients are stratified between high risk and low risk disease status.
  High risk patients receive 1 cycle of R-CODOX-M chemotherapy IV followed by R-IVAC chemotherapy over 30 minutes(Regimen B); regimens A and B are then repeated.
  Regimen A: Cyclophosphamide (800 mg/m2 IV over 1 hour)+ vincristine (1.5 mg/m2 IV PUSH)+ doxorubicin (40 mg/m2 IV)+ high-dose methotrexate (2,700 mg/m2 IV over 23 hours)+ rituximab (500 mg/m2 IV)(R-CODOX-M) regimen
- Low Risk - Treatment With 3 Cycles of R-CODOX-M: Patients are stratified between high risk and low risk disease status. Low risk patients receive 3 cycles of rituximab (500 mg/m2) R-CODOX-M chemotherapy IV over 2-4 hours with intrathecal chemotherapy (Regimen A).
  Regimen A: Cyclophosphamide (800 mg/m2 IV over 1 hour)+ vincristine (1.5 mg/m2 IV PUSH)+ doxorubicin (40 mg/m2 IV)+ high-dose methotrexate (2,700 mg/m2 IV over 23 hours)+ rituximab (500 mg/m2 IV)(R-CODOX-M) regimen
  Regimen B: Rituximab (500 mg/m2 IV once)+ Ifosfamide (1500 mg/m2 IV daily over 3 hours)+ Etoposide (60 mg/m2 IV daily over 1 hour), and Cytarabine (2 grams/m2 IV over 3 hours for 4 doses) 4 doses)
- Total: Total of all reporting groups
Arm/Group | High Risk - Treated With Alternating R-CODOX-M/R-IVAC Cycles | Low Risk - Treatment With 3 Cycles of R-CODOX-M | Total
Number analyzed (Participants) | 20 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 4 | 21
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 18 | 4 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 5 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 5 | 25
Human Immunodeficiency Virus (HIV) Status [Count of Participants; unit: Participants]
  Positive | 3 | 1 | 4
  Negative | 17 | 4 | 21
Lactate dehydrogenase (LDH) Level [Count of Participants; unit: Participants]
  Within Normal Range | 5 | 3 | 8
  Elevated | 15 | 2 | 17
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS) determines the ability of patients being able to tolerate therapies in serious illness. Scale is as follows:
  0 = Asymptomatic, normal activity
  1. = Symptomatic but completely ambulatory
  2. = Symptomatic, less than 50% of time in bed but not bedbound
  3. = In bed more than 50% of the time
  4. = 100% bedridden
  5. = death
  Participants
    0 | 8 | 1 | 9
    1 | 6 | 4 | 10
    2 | 6 | 0 | 6
Bulky disease [Count of Participants; unit: Participants] — Bulky disease is defined as disease in which there is a tumor mass more than 10 cm in its greatest diameter
  Participants
    Yes | 8 | 0 | 8
    No | 12 | 5 | 17
Ann Arbor Stage [Count of Participants; unit: Participants] — Classification for Hodgkin Lymphoma ranging from I-IV with IV being worse disease with liver or bone marrow, lungs or cerebrospinal fluid involvement.
  Participants
    Stage I | 1 | 3 | 4
    Stage II | 1 | 2 | 3
    Stage III | 3 | 0 | 3
    Stage IV | 15 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of Patients With Burkitt's and Burkitt-like Lymphoma/Leukemia Treated With Modified Magrath Regimen
Description: Response Rate is defined as combined number of patients with Complete Remission (CR) Complete Remission undetermined (Cru) and Partial Remission (PR) for patients with Burkitt's and Burkitt-like Lymphoma/Leukemia. Response will be measured by CT scans following treatment completion and assessed using Response Criteria for Non-Hodgkin's Lymphoma where:
  CR=complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms.
  CRu=same as above but allowing for 75% decrease in lymph node masses and indeterminate or normal bone marrow.
  PR=50% decrease in SPD of the six largest dominant nodes or nodal masses with no increase in size or other nodes, liver, spleen and no new sites of disease.
Time Frame: After two cycles of treatment and at completion of treatment (4 cycles for high risk and 3 cycles for low risk) up to approximately 20 weeks.
Population: One patient was determined not to be evaluable for response as he did not complete 2 cycles that were required per protocol to be evaluable for this outcome measure
Measure: Number; unit: percentage of patients
Groups:
- High Risk - Treated With Alternating R-CODOX-M/R-IVAC: Patients are stratified between high risk and low risk disease status.
  High risk patients receive 1 cycle of R-CODOX-M chemotherapy IV followed by R-IVAC chemotherapy over 30 minutes(Regimen B); regimens A and B are then repeated.
  Regimen A: Cyclophosphamide (800 mg/m2 IV over 1 hour)+ vincristine (1.5 mg/m2 IV PUSH)+ doxorubicin (40 mg/m2 IV)+ high-dose methotrexate (2,700 mg/m2 IV over 23 hours)+ rituximab (500 mg/m2 IV)(R-CODOX-M) regimen
  Regimen B: Rituximab (500 mg/m2 IV once)+ Ifosfamide (1500 mg/m2 IV daily over 3 hours)+ Etoposide (60 mg/m2 IV daily over 1 hour), and Cytarabine (2 grams/m2 IV over 3 hours for 4 doses)
Arm/Group | High Risk - Treated With Alternating R-CODOX-M/R-IVAC | Low Risk - Treatment With 3 Cycles of R-CODOX-M
Number analyzed (Participants) | 20 | 4
percentage of patients
  ORR after two cycles of treatment | 100 | 100
  ORR at completion of treatment | 100 | 100

2. Secondary Outcome: Overall Survival (OS) of Patients With Burkitt's and Burkitt-like Lymphoma/Leukemia Treated With Modified Magrath Regimen
Description: Overall Survival (OS) of patients with Burkitt's and Burkitt-like Lymphoma/Leukemia treated with modified Magrath regimen. OS is defined from the first dose of study drug to the time of death for any reason.
Time Frame: At 2 years from treatment initiation Median follow up 34 months (range 15-45)
Population: Evaluable patients for this outcome measure and were reported on together and in stratified group: high-risk and low-risk
Measure: Number; unit: percentage of patients alive
Arm/Group | High Risk - Treated With Alternating R-CODOX-M/R-IVAC | Low Risk - Treatment With 3 Cycles of R-CODOX-M
Number analyzed (Participants) | 20 | 4
percentage of patients alive | 81 | 100

3. Secondary Outcome: Safety of Patients With Burkitt's and Burkitt-like Lymphoma/Leukemia Treated With Modified Magrath Regimen (Addition of Rituximab, Subsitution of Adriamycin for Doxil and Using Lower Dose of Methotrexate)
Description: Adverse events (AE) graded as either 3 or 4 and determined to be at least possibly related to study treatment will be collected in patients Burkitt's and Burkitt-like Lymphoma/Leukemia treated with modified Magrath regimen to assess the safety and toxicity profile of the addition of rituximab, subsitution of adriamycin for doxil and lower dose of methotrexate. AEs will be assessed as follows at the following time points: At the end of each cycle or monthly whichever is less frequent and 30 days post last dose of study treatment for a maximum of 3 cycles for regimen A and 4 cycles for regimen B and up to 12 months.
  In general AEs will be assessed according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v 3.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: After each cycle or monthly (whichever is less frequent), 30 days post last dose. Treatment duration was at a median of 13 weeks (range 11-20) for high-risk patients and 10 weeks (range 9-12) for low-risk patients.
Population: All patients that receive at least one dose of study drug are evaluable for this outcome measure
Measure: Number; unit: participants
Arm/Group | High Risk - Treated With Alternating R-CODOX-M/R-IVAC | Low Risk - Treatment With 3 Cycles of R-CODOX-M
Number analyzed (Participants) | 20 | 5
participants
  Anemia : Grade 3 | 13 | 3
  Anemia : Grade 4 | 1 | 0
  Neutropenia : Grade 3 | 5 | 2
  Neutropenia : Grade 4 | 6 | 2
  Thrombocytopenia : Grade 3 | 1 | 1
  Thrombocytopenia : Grade 4 | 13 | 2
  Mucositis : Grade 3 | 7 | 2
  Mucositis : Grade 4 | 3 | 0
  Infection : Grade 3 | 8 | 1
  Infection : Grade 4 | 0 | 0
  Elevated Transaminases : Grade 3 | 6 | 2
  Elevated Transaminases : Grade 4 | 0 | 0
  Fever (Neutropenic) : Grade 3 | 4 | 3
  Fever (Neutropenic) : Grade 4 | 0 | 0
  Low Phosphate : Grade 3 | 5 | 1
  Low Phosphate : Grade 4 | 0 | 0
  Sodium Abnormalities : Grade 3 | 4 | 2
  Sodium Abnormalities : Grade 4 | 0 | 0
  Hyperglycemia : Grade 3 | 1 | 3
  Hyperglycemia : Grade 4 | 5 | 0
  Hypoalbuminemia : Grade 3 | 4 | 0
  Hypoalbuminemia : Grade 4 | 0 | 0
  Hypokalemia : Grade 3 | 1 | 2
  Hypokalemia : Grade 4 | 0 | 0
  Cardiac : Grade 3 | 3 | 0
  Cardiac : Grade 4 | 0 | 0
  Diarrhea : Grade 3 | 2 | 0
  Diarrhea : Grade 4 | 0 | 0
  Elevated Creatinine : Grade 3 | 2 | 0
  Elevated Creatinine : Grade 4 | 0 | 0
  Nausea/Vomiting : Grade 3 | 1 | 0
  Nausea/Vomiting : Grade 4 | 0 | 0
  Low Blood Pressure : Grade 3 | 1 | 0
  Low Blood Pressure : Grade 4 | 0 | 0
  Rash : Grade 3 | 1 | 0
  Rash : Grade 4 | 0 | 0
  Edema : Grade 3 | 1 | 0
  Edema : Grade 4 | 0 | 0
  Low Magnesium : Grade 3 | 1 | 0
  Low Magnesium : Grade 4 | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS) of Patients With Burkitt's and Burkitt-like Lymphoma/Leukemia Treated With Modified Magrath Regimen
Description: Progression Free Survival (PFS) will be defined from the first dose of study drug to the first documentation of progressive disease or death for any reason. Patients that are lost to follow-up before progression will be censored at the point of last documentation of not experiencing the event.
Time Frame: At 2 years from treatment initiation. Median follow up 34 months (range 15-45)
Population: as for outcome 2
Measure: Number; unit: percentage of patients progression free
Arm/Group | High Risk - Treated With Alternating R-CODOX-M/R-IVAC | Low Risk - Treatment With 3 Cycles of R-CODOX-M
Number analyzed (Participants) | 20 | 4
percentage of patients progression free | 76 | 100

ADVERSE EVENTS:
Time Frame: Safety data was collected on Day 1 of each cycle of chemotherapy, for the previous cycle or monthly, whichever was less frequent and 30 days post last dose of study treatment. Treatment duration was at a median of 13 weeks (range 11-20) for high-risk patients and 10 weeks (range 9-12) for low-risk patients.
Groups:
- High Risk - Treated With Alternating R-CODOX-M/R-IVAC Cycles: Patients are stratified between high risk and low risk disease status.
  High risk patients receive 1 cycle of R-CODOX-M chemotherapy IV followed by R-IVAC chemotherapy over 30 minutes(Regimen B); regimens A and B are then repeated.
  Regimen A: Cyclophosphamide (800 mg/m2 IV over 1 hour)+ vincristine (1.5 mg/m2 IV PUSH)+ doxorubicin (40 mg/m2 IV)+ high-dose methotrexate (2,700 mg/m2 IV over 23 hours)+ rituximab (500 mg/m2 IV)(R-CODOX-M) regimen
  Regimen B: Rituximab (500 mg/m2 IV once)+ Ifosfamide (1500 mg/m2 IV daily over 3 hours)+ Etoposide (60 mg/m2 IV daily over 1 hour), and Cytarabine (2 grams/m2 IV over 3 hours for 4 doses)
Arm/Group | High Risk - Treated With Alternating R-CODOX-M/R-IVAC Cycles | Low Risk - Treatment With 3 Cycles of R-CODOX-M
All-Cause Mortality (participants affected / at risk) | 4/20 | 0/5
Serious Adverse Events (participants affected / at risk) | 20/20 | 2/5
Other Adverse Events (participants affected / at risk) | 20/20 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk - Treated With Alternating R-CODOX-M/R-IVAC Cycles (N=20) | Low Risk - Treatment With 3 Cycles of R-CODOX-M (N=5)
myelodysplastic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Systematic Assessment
Cardiac dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Pleuritic chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Cerebritis (General disorders) | 1 (1) | 0 (0)
Febrile neutropnia (Infections and infestations) | 5 (7) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Bloodinfection (Infections and infestations) | 1 (1) | 0 (0)
Pancytopenia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Neuro symptoms - Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Renal failuretumor lysis syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk - Treated With Alternating R-CODOX-M/R-IVAC Cycles (N=20) | Low Risk - Treatment With 3 Cycles of R-CODOX-M (N=5)
Allergic reaction/ hypersensitivity (including drug fever) (Immune system disorders) | 1 | 0
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 18 | 5
Neutrophils (neutropenia) (Blood and lymphatic system disorders) | 11 | 3
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 20 | 5
Lymphopenia (Blood and lymphatic system disorders) | 10 | 3
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 20 | 4
Hypertension (Cardiac disorders) | 5 | 1
Hypotension (Cardiac disorders) | 4 | 1
Cardiac General (Cardiac disorders) | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 2 | 1
LVEF (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 18 | 2
Fever (General disorders) | 4 | 2
Rigors (General disorders) | 1 | 0
Sweating (General disorders) | 1 | 0
Weight loss (General disorders) | 6 | 2
Weight gain (General disorders) | 1 | 0
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 | 0
Brusing (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 8 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 | 0
Anorexia (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 3
Colitis (Gastrointestinal disorders) | 1 | 0
Dehydration (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 10 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 0
GI obstruction (Gastrointestinal disorders) | 1 | 0
Mucositis/stomatitis (Gastrointestinal disorders) | 18 | 4
Nausea (Gastrointestinal disorders) | 12 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1
Stomach Pain (Gastrointestinal disorders) | 1 | 0
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 11 | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 0
Bleeding gums (Skin and subcutaneous tissue disorders) | 1 | 0
Nose bleed (General disorders) | 1 | 1
Febrile neutropenia (Infections and infestations) | 8 | 3
Colitis, infectious (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Abdomen infection (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Rash (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Infection NOS (Infections and infestations) | 1 | 0
Infected ommaya (Infections and infestations) | 1 | 0
Edema:limb (Blood and lymphatic system disorders) | 5 | 0
Edema:head and neck (Blood and lymphatic system disorders) | 3 | 0
Alkaline phosphatase (Metabolism and nutrition disorders) | 12 | 3
Transaminase increased (Metabolism and nutrition disorders) | 14 | 3
ALT, SGPT (serum glutamic pyruvic transaminase) atinine (Metabolism and nutrition disorders) | 4 | 2
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 12 | 2
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 8 | 3
Bicarbonate - low (Metabolism and nutrition disorders) | 5 | 2
Creatinine increased (Metabolism and nutrition disorders) | 7 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 13 | 3
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 2 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 18 | 5
Glucose, serum-low(hypoglycemia) (Metabolism and nutrition disorders) | 4 | 0
Lactic acid dehydrogenase (LDH) increase (Metabolism and nutrition disorders) | 1 | 0
Magnesium, serum-low(hypomagnesemia) (Metabolism and nutrition disorders) | 10 | 0
Phosphate, serum-high (hyperphosphatemia) (Metabolism and nutrition disorders) | 0 | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 9 | 0
Potassium, serum-low(hypokalemia) (Metabolism and nutrition disorders) | 14 | 2
Sodium, serum-high(hypernatremia) (Metabolism and nutrition disorders) | 2 | 0
Sodium, serum-low(hyponatremia) (Metabolism and nutrition disorders) | 12 | 2
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 5 | 1
Neuropathy: motor (Nervous system disorders) | 1 | 0
Foot drop (Motor Neuopathy) (Nervous system disorders) | 1 | 0
Neuropathy:sensory (Nervous system disorders) | 6 | 1
Dizziness (Psychiatric disorders) | 1 | 1
Memory impairment (Psychiatric disorders) | 1 | 0
Mood alteration - Anxiety (Psychiatric disorders) | 1 | 0
Mood alteration - Depression (Psychiatric disorders) | 0 | 1
Nerve pain (Nervous system disorders) | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) Whole body/generalized (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in throat (Gastrointestinal disorders) | 1 | 0
Pain in abdomen NOS (Gastrointestinal disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in esophagus (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Epigastrium (Musculoskeletal and connective tissue disorders) | 1 | 0
Oral pain (General disorders) | 7 | 1
Peri-rectal pain (General disorders) | 0 | 1
Head/headache (Nervous system disorders) | 9 | 3
Pain NOS (General disorders) | 7 | 1
Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Carbon monoxide diffusion capacity (DLCO) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Floaters (Eye disorders) | 1 | 0
Double vision (Eye disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 1
Urinary frequency retention (Renal and urinary disorders) | 1 | 0
Obstrution (Renal and urinary disorders) | 1 | 0
Flu-like syndrome (General disorders) | 1 | 0
Vision photophobia (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes